CLINICAL TRIAL: NCT02383901
Title: A Retrospective Non-intervention Study to Characterize FOlate Rescue Treatment in Osteosarcoma Patients Treated With HDMTX
Acronym: FORTO
Status: Completed | Type: Observational
Sponsor: Isofol Medical AB (Industry)
Responsible Party: Sponsor
Other Study IDs: ISO-MTX-OB1
Record Dates: First submitted 2014-10-29; First posted 2015-03-10 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — Methotrexate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Methotrexate — The study includes osteosarcoma patients who have received MAP treatment, MAP treatment contains 12 courses of Methotrexate

SUMMARY:
The purpose of this study is to investigate to which extend osteosarcoma patients do NOT meet the criteria for successfully advancement to next planned chemotherapy course.

DETAILED DESCRIPTION:
Methotrexate is one of the most effective chemotherapy drugs in the treatment of osteosarcoma. However, it has severe side effects. The physicians tries to save or "rescue" normal cells from the side effects of methotrexate by giving folinic acid. Folinic acid administration starts 24 hours after methotrexate and given regularly until methotrexate levels are low and not dangerous to normal cells anymore. Despite this rescue, side effects are still a problem and many patients are not well enough to receive subsequent chemotherapy on time.

This is a multi-center, observational retrospective study with osteosarcoma patients, 2 years of age or older, who have received at least one (1) course of HDMTX treatment with folate rescue in a MAP schedule between 01January 2009 and 31 May 2014, both dates included.

Patients must have initiated their HDMTX treatment after 01 January 2009, received at least one (1) course of HDMTX treatment with folate rescue, and received their last MAP intervention (regardless if the patients received all planned HDMTX treatments or terminated prematurely their treatment) by 31 May 2014.

Patient data collected for the study will be extracted from hospital medical records and will include information related to scheduled and/or received HDMTX courses. The collected data will include: laboratory values confirming suitability to receive next chemotherapy intervention at scheduled time, drug administration regimen (both HDMTX and supportive care), toxicity management (hydration and folate rescue regimens), and toxicity monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological evidence of osteosarcoma including metastatic osteosarcoma.
* Patients must have initiated their HDMTX treatment after 01 January 2009 and should have completed their MAP treatment by 31 May 2014.
* Patients should have received at least one (1) HDMTX course within MAP treatment.
* Patients must be at least 2 years of age.
* Patient, parent(s), or guardian(s), as appropriate, is/are willing to provide signed informed consent, if applicable according to national regulation.

Exclusion Criteria:

* No exclusion criteria

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Osteosarcoma patients, 2 years of age or older. Patients must have received at least one course of HDMTX treatment with folate rescue in a MAP schedule. The treatment must have been initiated by 01 January 2009 and completed by 31 May, 2014
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients classified as NOT having met the criteria for successful advancement from the first to second HDMTX course within the same MAP and/or next MAP cycle at scheduled time in any given HDMTX courses. | Druing the MAP treatment approx 30 weeks

SECONDARY OUTCOMES:
Administrated HDMTX courses classified as NOT having met the criteria for successful advancement from first to second HDMTX course and/or from the second HDMTX course to the next MAP cycle at scheduled time. | Druing the MAP treatment approx 30 weeks
Number of patients with MTX excretion toxicity | Druing the MAP treatment approx 30 weeks
AEs and laboratory test values that resulted in change of folate management reported during the MAP cycle that led or contributed to NOT successfully advancement to next treatment at scheduled time. | Druing the MAP treatment approx 30 weeks
AEs and laboratory test values reported during the MAP cycle that led or contributed to changes in planned hydration strategy. | Druing the MAP treatment approx 30 weeks
AEs and laboratory test values reported during the MAP cycle that led or contributed to changes in planned folate rescue strategy. | Druing the MAP treatment approx 30 weeks
Characterization of the S-MTX elimination profile and management | Druing the MAP treatment approx 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Eriksson, MD PhD., Principal Investigator — Skåne Universitiy Hospital
Locations (5):
- Semmelweis Egyetem II. Sz. Gyermekklinika, Budapest, Hungary
- Oslo University Hospital, Oslo, Norway
- Intytut Matki Dziecka Klinika Chirurgii Onkologicznej Dzieci i Młodzieży, Warsaw, Poland
- Sweden (2):
  - Skåne University Hospital, Lund
  - Karolinska University Hospital, Sweden, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Publication in relevant forum planned after finalization of study report